CLINICAL TRIAL: NCT00703755
Title: A Randomized, Double-Blind Trial Comparing the Efficacy and Safety of Fenofibrate, Metformin, Their Combination and Placebo in Patients With Metabolic Syndrome.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Bruno Fraitag, Solvay Pharmaceuticals
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: CFEN0203
Record Dates: First submitted 2008-06-20; First posted 2008-06-23 (Estimated); Last update posted 2008-06-25 (Estimated); Status verified 2008-06

CONDITIONS: Patients With Metabolic Syndrome
Keywords: Diabetes; Hypertriglyceridaemia; Metabolic Syndrome
MeSH Terms: conditions — Diabetes Mellitus; Hypertriglyceridemia; Metabolic Syndrome | interventions — Fenofibrate; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- 1 (Experimental)
  Interventions: Drug: Fenofibrate /Metformin
- 2 (Experimental)
  Interventions: Drug: Fenofibrate /Metformin
- 3 (Experimental)
  Interventions: Drug: Fenofibrate /Metformin
- 4 (Experimental)
  Interventions: Drug: Fenofibrate /Metformin
- 5 (Experimental)
  Interventions: Drug: Fenofibrate /Metformin
- 6 (Experimental)
  Interventions: Drug: Fenofibrate /Metformin
- 7 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fenofibrate /Metformin — fenofibrate 2 x 40 mg bid + metformin 850 mg bid (F160-M1700)
  Arms: 1
Drug: Fenofibrate /Metformin — fenofibrate 2 x 40 mg bid + metformin 500 mg bid (F160-M1000)
  Arms: 2
Drug: Fenofibrate /Metformin — fenofibrate 40 mg bid + metformin 850 mg bid (F80-M1700)
  Arms: 3
Drug: Fenofibrate /Metformin — fenofibrate 40 mg bid + metformin 500 mg bid (F80-M1000)
  Arms: 4
Drug: Fenofibrate /Metformin — fenofibrate 2 x 40 mg bid + metformin placebo (F160-M0)
  Arms: 5
Drug: Fenofibrate /Metformin — fenofibrate placebo + metformin 850 mg bid (F0-M1700)
  Arms: 6
Drug: Placebo — Placebo
  Arms: 7

SUMMARY:
The purpose of this study was to study the effect of different combinations of fenofibrate and metformin on the cluster of metabolic syndrome (MetS) biochemical abnormalities, and to determine the dose combination allowing normalization of MetS patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged from 18 to 75 years old (at inclusion V1).
* With 3 of the following 5 criteria, including at least 2 biochemical abnormalities (glucose and one lipid abnormality)
* And having signed a written informed consent (at inclusion V1).

Exclusion Criteria:

* known Type 1 diabetes, or treated type 2 diabetes [25], [26];
* wth HbA1c > 8 % [27] at the first blood sample;
* body mass index (BMI) > 45 kg/m2;
* females who were not surgically sterilized or not using adequate contraceptive or not using adequate contraceptive precautions or not postmenopausal
* pregnant or lactating women;
* known hypersensitivity to fibrates;
* known hypersensitivity to metformin chlorhydrate; known abnormal thyroid hormone levels, or high thyroid stimulating hormone (TSH) level;
* having received an investigational drug in the last 30 days before the date of randomization;
* unable or unwilling to comply with the protocol;
* likely to withdraw from the study before its completion;
* treated with some concomitant medications:
* reporting a change within the last 6 weeks before randomization and during the study in the medications that could interfere with the lipid profile (i.e., anti-hypertensive drugs, oral corticosteroids, thyroid hormones, retinoids, thiazidic derivatives, hormone replacement therapies);
* presenting with the following disease or conditions:

  * chronic respiratory insufficiency, patient with medical device for sleep apnea;
  * current chronic pancreatitis, or identified risk or known history of acute pancreatitis;
  * hepatic insufficiency, acute alcohol intoxication, alcoholism;
  * known cholelithiasis without cholecystectomy;
  * aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 2 times the upper limit normal (ULN);
  * musculoskeletal disease or increased creatine phosphokinase (CPK) > 3 times the ULN;
  * renal failure or renal dysfunction defined by serum creatinine levels > 135 μmol/L in males and > 110 μmol/L in females [28];
  * acute conditions with the potential to alter renal function such as dehydration, severe infection, shock or intravascular administration of iodinated contrast agents;
  * acute or chronic disease which may cause tissue hypoxia such as cardiac or respiratory failure, recent myocardial infarction (within 3 months prior to randomization), shock;
  * known gastric or peptic ulcer or intestinal disease within the previous 3 months of randomization capable of modifying the intestinal absorption of the drugs;
  * any other severe pathology such as cancer, mental illness, etc., which in the opinion of the investigator might pose a risk to the patient or confound the results of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2288 (Actual)
Dates: Start 2003-03; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
The percentage of normalized patients at V4 (fasting glucose < 6.1 mmol/L, TG < 1.69 mmol/L and HDL-C >= 1.03 mmol/L in males and >= 1.29 mmol/L in females) | End of study visit (V4)

SECONDARY OUTCOMES:
Fasting blood insulin and fasting blood glucose, HbA1c. | End of study visit (V4)
Area under the curve from 0 to 2h (AUC0-2h) of glucose, insulin, C-peptide and free fatty acids (FFA) during Oral Glucose Tolerance Test (OGTT). | End of study visit (V4)
Insulin sensitivity assessed by the OGTT-derived composite whole-body Insulin Sensitivity Index (ISI) | End of study visit (V4)
Fasting lipid parameters: FFA, TG, TC, HDL-C, measured LDL-C, VLDL-C, small dense LDL, apolipoprotein (Apo) A1, Apo A2, Apo CIII, LDL and HDL sizes, remna | End of study visit (V4)
Plasminogen -1 Activation Inhibitor (PAI-1) activity, PAI-1 antigen, tissue-type Plasminogen Activator antigen (t-PA-ag), high sensitivity C-reactive protein (hsCRP), fibrinogen, tumor necrosing factor (TNF) alpha, interleukin (IL)1 and IL6. | End of study visit (V4)
Body mass index (BMI), waist circumference, hip circumference, waist to hip ratio, and blood pressure. | End of study visit (V4)
Percentage of patients who presented 0, 1, 2, 3, 4 or 5 MetS criteria. | End of study visit (V4)
Adverse events (AEs). | End of study visit (V4)
Biochemistry: creatinine phosphokinase (CPK), AST, ALT, GGT, alkaline phosphatase, serum creatinine, total bilirubin, blood urea nitrogen (BUN), uric acid, albumin and total homocysteine | End of study visit (V4)
Hematology: white blood cells (WBC) and differential count, red blood cells (RBC), hemoglobin, hematocrit and platelets. | End of study visit (V4)
Blood pressure. | End of study visit (V4)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (101):
- Canada (21):
  - Site 013, Calgary, Alberta
  - Site 019, Calgary, Alberta
  - Site 007, Chicoutimi
  - Site 024, Halifax
  - Site 004, Hamilton
  - Site 012, Kingston
  - Site 017, Longueuil
  - Site 009, Montague
  - Site 001, Montreal
  - Site 015, Montreal
  - Site 003, Québec
  - Site 025, Sainte-Foy
  - Site 026, Sainte-Foy
  - Site 021, Sherbrooke
  - Site 010, St. John's
  - Site 020, St. John's
  - Site 022, St. John's
  - Site 006, Ste-Foy
  - Site 016, Toronto
  - Site 005, Vancouver
  - Site 011, Victoria
- Finland (6):
  - Site 090, Hus
  - Site 091, Jakobstad
  - Site 095, Jyväskylä
  - Site 092, Mikkeli
  - Site 096, Närpes
  - Site 094, Vaasa
- Hungary (16):
  - Site 190, Budapest
  - Site 191, Budapest
  - Site 193, Budapest
  - Site 199, Budapest
  - Site 202, Budapest
  - Site 204, Budapest
  - Site 203, Debrecen
  - Site 200, Gyöngyös
  - Site 201, Győr
  - Site 198, Gyula
  - Site 197, Miskolc
  - Site 196, Pécs
  - Site 194, Szeged
  - Site 192, Székesfehérvár
  - Site 205, Szombathely
  - Site 195, Veszprém
- Italy (7):
  - Site 074, Catanzaro
  - Site 077, Chieti Scalo
  - Site 075, Padua
  - Site 076, Padua
  - Site 073, Palermo
  - Site 072, Perugia
  - Site 070, Treviglio Bergamo
- Netherlands (18):
  - Site 044, Almere Stad
  - Site 040, Amsterdam-Zuidoost
  - Site 054, Den Helder
  - Site 057, Dordrecht
  - Site 042, Eindhoven
  - Site 045, Groningen
  - Site 052, Groningen
  - Site 041, Hoorn
  - Site 046, Leiden
  - Site 047, Rotterdam
  - Site 051, Rotterdam
  - Site 043, Sliedrecht
  - Site 055, Tiel
  - Site 053, Veldhoven
  - Site 048, Velp
  - Site 056, Velp
  - Site 049, Zoetermeer
  - Site 060, Zwijndrecht
- Norway (8):
  - Site 117, Elverum
  - Site 114, Hobol
  - Site 111, Horten
  - Site 110, Oslo
  - Site 112, Oslo
  - Site 113, Oslo
  - Site 118, Oslo
  - Site 115, Skedsmokorset
- Poland (8):
  - Site 130, Brodnowski
  - Site 139, Chrzanów
  - Site 134, Gdansk
  - Site 132, Katowice
  - Site 131, Kielce
  - Site 135, Olsztyn
  - Site 138, Ul. Ziolowa
  - Site 133, Warsaw
- Romania (11):
  - Site 220, Brasov
  - Site 210, Bucharest
  - Site 211, Bucharest
  - Site 212, Bucharest
  - Site 214, Bucharest
  - Site 218, Bucharest
  - Site 219, Bucharest
  - Site 215, Cluj-Napoca
  - Site 213, Craiova
  - Site 217, Iași
  - Site 216, Suceava
- Sweden (6):
  - Site 153, Gothenburg
  - Site 154, Kristianstad
  - Site 150, Linköping
  - Site 155, Lund
  - Site 152, Stockholm
  - Site 151, Umeå